CLINICAL TRIAL: NCT05918601
Title: Effectiveness of a Peer-led Personalized Support Program Using Instant Messaging Applications and a Self-determination Theory-based Intervention to Help Young Drug Abusers Quit Drugs: A Randomized Controlled Trial
Brief Title: Peer-led Personalized Support Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Li Ho Cheung William, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NTEC-2023-129
Record Dates: First submitted 2023-04-13; First posted 2023-06-26 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Health-risk Behaviours; Drug Abuse
Keywords: Health-risk Behaviours; Drug Abuse
MeSH Terms: conditions — Substance-Related Disorders | interventions — Theory of Planned Behavior; Models, Biological; Videotape Recording

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Each participant will receive the telephone that will be delivered by a trained peer supporter using the Ask, Warn, Advise, Refer and Do-it-Again (AWARD) model. For the advice steps, participants will be asked about the priority they place on engagement in health-related lifestyles. A brief intervention on the selected health-related lifestyle will be given. In addition, they will be informed that they will receive instant messaging via WeChat or WhatsApp to assist them to adhere to their schedule of the desirable health-related lifestyle throughout the study period. For the first 6 months of the study period, peer supporters will send WhatsApp or WeChat messages approximately once per week to the participants to remind them to adhere to their schedule of the desirable health-related lifestyle. In addition, the participants will receive four independent 1-minute videos which focus on the health risks associated with abusing drugs and the benefits of quitting drugs.
  Interventions: Other: Health-risk behaviors; Other: Theory of planned behavior, Self-determination theory; Other: Assist them to adhere to their schedule of quitting drugs throughout the study period; Other: Assist them to adhere to their schedule of desirable health-related lifestyles/quitting drugs throughout the study period; Other: (AWARD) model; Other: Receive four independent 1-minute videos
- Control Group (Placebo Comparator): Trained peer supporters will answer calls from potential participants and explain the nature and purpose of the project to them. Each participant will then receive a brief intervention over the telephone that will be delivered by a trained peer supporter using the Ask, Warn, Advise, Refer and Do-it-Again (AWARD) model. Participants will be asked to quit drugs immediately or progressively. In addition, they will be informed that they will receive instant messaging via WeChat or WhatsApp from peer supporters to assist them to adhere to their schedule of quitting drugs throughout the study period. For the first six months, participants will receive four independent 1-minute videos which focus on the health risks associated with abusing drugs and the benefits of quitting drugs without any schedule of the desirable health-related lifestyle throughout the study period.
  Interventions: Other: Theory of planned behavior, Self-determination theory; Other: Assist them to adhere to their schedule of quitting drugs throughout the study period; Other: (AWARD) model; Other: Receive four independent 1-minute videos

INTERVENTIONS:
Other: Health-risk behaviors — Participants will be asked about the priority they place on engagement in health-related lifestyles, such as quitting drugs, alcohol, smoking or exercising regularly.
  Arms: Intervention group
Other: Theory of planned behavior, Self-determination theory — The participants will be asked to quit drugs immediately or progressively with the ultimate goal of quitting drugs completely.
Other: Assist them to adhere to their schedule of quitting drugs throughout the study period — The participants will receive instant messaging via WeChat or WhatsApp from peer supporters to assist them to adhere to their schedule of quitting drugs throughout the study period.
Other: Assist them to adhere to their schedule of desirable health-related lifestyles/quitting drugs throughout the study period — The participants will receive instant messaging via WeChat or WhatsApp from peer supporters to assist them to adhere to their schedule of desirable health-related lifestyles/quitting drugs throughout the study period.
  Arms: Intervention group
Other: (AWARD) model — Participants receive a brief intervention using the Ask, Warn, Advise, Refer and Do-it-Again (AWARD) model
Other: Receive four independent 1-minute videos — The participants will receive four independent 1-minute videos which focus on the health risks associated with abusing drugs and the benefits of quitting drugs.

SUMMARY:
Aim: To test the effectiveness of a peer-led personalized support program using instant messaging applications and a self- determination theory-based intervention to help young drug abusers quit drugs.

Hypothesis to be tested: The investigators hypothesize that compared with those in the control group, the participants in the intervention group will experience greater success in reducing and quitting drugs and will have a better health-related quality of life at 12 months follow-up.

DETAILED DESCRIPTION:
Setting:

A pre- and post-test interventional study will be conducted in the peer supporters. A randomized controlled trial (RCT) will be carried out attaching to this service to evaluate the effects of engagement in the desirable health-related lifestyle on the drug quitting of adolescent drug abusers in Hong Kong.

There will be a target drug abusers service group and peer supporters group. It is expected that the project will receive 1,000 telephone inquiries and provide phone drug abstinence intervention to about 200 drug-abusing youths or young adults and randomized into two groups (100 eligible participants in intervention and eligible 100 participants in control group) and recruit about 80 university students as peer supporters.

To raise anti-drug awareness among young people and identify high-risk/hidden drug-abusing young people aged 35 or below in Hong Kong, there are at least 30,000 pamphlets, booklets and other publicity materials will be delivered to students and teachers at secondary schools and tertiary institutions, to young members of youth organisations and to young employees in high-pressure industries. Approximately 200 secondary and tertiary schools, 50 youth organisations and 50 companies in high-pressure industries will be targeted to introduce the peer-led personalised support programme to teachers, school social workers, students, and young employees and organisation members.

To train university students with medical backgrounds to become peer-led personalised supporters who will implement a brief intervention and provide continual personalised support to help young drug abusers quit drugs.

To implement a peer-led personalised support programme to help young drug abusers quit drugs by using instant messaging applications and a self-determination theory-based intervention

Intervention:

Each participant will then receive a brief intervention over the telephone that will be delivered by a trained peer supporter using the Ask, Warn, Advise, Refer and Do-it-Again (AWARD) model, which was originally developed for primary-care tobacco-cessation interventions. The brief intervention will include the following steps: (1) ask about and assess drug abuse history; (2) warn about the health hazards associated with such health-risk behaviour; (3) advise on how to quit drugs; (4) refer to drug rehabilitation organisations for quitting drugs on request and (5) repeat steps 1 to 4. Participants will be asked about the priority participants place on engagement in health-related lifestyles, such as quitting drugs, alcohol, smoking or exercising regularly. A brief intervention on the selected health-related lifestyle will be given. In addition, participants will be informed that participants will receive instant messaging via WeChat or WhatsApp from peer supporters to assist drug abusers to adhere to schedule of the desirable health-related lifestyle throughout the study period. The duration of the entire intervention will be approximately 5-10 minutes but will be slightly longer if necessary. Such a brief intervention will be cost-effective and more feasible than other interventions for routine use by peer supporters after minimal training. Previous clinical trials of smoking cessation have provided strong evidence on the effectiveness of brief interventions using the AWARD model.

For the first 6 months of the study period, peer supporters will send WhatsApp or WeChat messages approximately once per week to the participants to remind the participants to adhere to schedule of the desirable health-related lifestyle. These messages will be delivered more often, if preferred by the participants. In addition, the participants will receive four independent 1-minute videos (one video will be sent in weeks 1, 5, 12 and 24, respectively) via WhatsApp or WeChat. The video content will focus on the health risks associated with abusing drugs and the benefits of quitting drugs. Participants will be assessed at 1 week, 1 month, 3 months, 6 months, 9 months and 12 months via telephone call. For those participants who have an intention of quitting drugs, participants will be allowed to select preferred quit schedules (quit immediately, or quit progressively, with the ultimate goal of quitting drugs completely).

After 6 months and until 12 months of follow-up, minimal messages will be sent by the peer supporters. These messages will enable the participants' progress to be followed and participants' questions to be answered, and maintain contact with the participants.

Control Group:

Trained peer supporters will answer calls from potential participants and explain the nature and purpose of the project to potential participants. Verbal consent to participate in the project will then be sought from eligible drug abusers. In addition, demographic and baseline data will be obtained. Each participant will then receive a brief intervention over the telephone that will be delivered by a trained peer supporter using the Ask, Warn, Advise, Refer and Do-it-Again (AWARD) model, which was originally developed for primary-care tobacco-cessation interventions. The brief intervention will include the following steps: (1) ask about and assess drug abuse history; (2) warn about the health hazards associated with such health-risk behaviour; (3) advise on how to quit drugs; (4) refer to drug rehabilitation organisations for quitting drugs on request and (5) repeat steps 1 to 4. Participants will be asked to quit drugs immediately or progressively. In addition, participants will be informed that participants will receive instant messaging via WeChat or WhatsApp from peer supporters to assist participants to adhere to schedule of quitting drugs throughout the study period.

For the first 6 months of the study period, peer supporters will send WhatsApp or WeChat messages approximately once per week to the participants to remind participants to adhere to schedule of quitting drugs. These messages will be delivered more often, if preferred by the participants. In addition, the participants will receive four independent 1-minute videos (one video will be sent in weeks 1, 5, 12 and 24, respectively) via WhatsApp or WeChat. The video content will focus on the health risks associated with abusing drugs and the benefits of quitting drugs. Participants will be assessed at 1 week, 1 month, 3 months, 6 months, 9 months and 12 months via telephone call to determine the participants' success in quitting drugs.

After 6 months and until 12 months of follow-up, minimal messages will be sent by the peer supporters. These messages will enable the participants' progress to be followed and participants' questions to be answered, and maintain contact with the participants.

Instruments:

A telephone record sheet will be used to record the incoming telephone calls. Both worldwide validated and self-administered measures (constructed based on previous studies of the PI & Co-Is and other worldwide validated measures) will be applied in the programme. Callers will be invited to complete a telephone interview in each of the telephone counselling (at baseline, 1-week, 1-month, 3-month, 6-month, 9-month, 12-month). The questionnaire assesses (a) drug abuse profile (quit history, no. of days use, daily drug consumption, etc), (b) drug dependency, (c) contemplation stage of drug abuse abstinence, (d) risk for relapsing, (e) quality of life, (f) withdrawal symptoms, (g) other health-related lifestyles and Demographics will also be asked during the baseline phone interview.

Subject recruitment :

The details of the nature and purpose of the project will be posted at website, secondary schools and tertiary institutions, youth organisations or NGOs, social platform and companies in high-pressure industries to identify potential participants. Young drug abusers will be able to express willingness to join the project by calling the telephone hotline provided. The hotline service will operate from 5 p.m. to 9 p.m. on weekday and from 2 p.m. to 8 p.m. on weekend. A peer supporter or a research assistant will answer the telephone inquiries from 9:00 a.m. to 5 p.m. on weekdays. Voice mails will be recorded during non-operating hours and public holidays. The hotline centre will close in case of bad weather (e.g. black rainstorm, hoisting of tropical cyclone signal No. 8).

Methods of Statistical Analysis:

Data will be entered and analyzed using IBM SPSS Statistics for Windows or R language programme. A significance level of 0.05 will be adopted. Following the Russell standard, intention-to-treat analysis will performed with the assumption that all participants lost to follow-up had no changes with the status at baseline. All missing data will be handled using multiple imputation.

Descriptive statistics such as frequency, percentage, Chi-square test and/or t-test will be used to measure the outcomes such as reduction of drug abuse consumption and other variables. Longitudinal repeated analysis will be used to measure the trend of drug reduction and other secondary outcome. Exploring subgroup analyses and sensitivity analysis will be performed.

ELIGIBILITY:
The inclusion criteria of target service group (drug abusers) for this programme:

* be aged 35 or below
* be able to communicate in Cantonese
* have an history of drug abuse within the past 12 months (including all types of drugs such as narcotics analgesics, hallucinogens, depressants, stimulants, tranquillizers and other recreational drugs)

The exclusion Criteria of target service group (drug abusers) for this programme:

* psychologically or physically unable to communicate

The inclusion criteria of peer supporters:

* be aged 18 - 35
* be able to communicate in Cantonese
* have a medical background
* complete the training courses and pass the evaluation of peer supporter qualification

The exclusion Criteria of peer supporters:

* psychologically or physically unable to communicate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Drug Consumption | 12 month
  Participants' change in drug consumption between baseline and 12-month follow-up will be measured by a structured-questionnaire. The questionnaire gathers the frequency and categories of drug consumption in the past 30 days. The more frequencies and the more kinds of drug used indicating the higher consumption of drug abuse.

SECONDARY OUTCOMES:
The self-reported drug abuse abstinence rate | 6 month and 12 month
  Participants' drug abuse abstinence between baseline, 6-month follow-up and 12-month follow-up will be measured by a structured-questionnaire. The questionnaire gathers the self-reported drug abuse abstinence in the past 30 days (do not use drug for at least 30 days during the time of follow-up).
The change in drug consumption | 6 month
  Participants' change in drug consumption between baseline and 6-month follow-up will be measured by a structured-questionnaire. The questionnaire gathers the frequency and categories of drug consumption in the past 30 days. The more frequencies and the more kinds of drug used indicating the higher consumption of drug abuse.
The changes of the contemplation stages at 6-month and 12-month | 6 month and 12 month
  Participants' changes of the contemplation stages between baseline, 6-month and 12-month follow-up will be measured by a structured-questionnaire of Contemplation Ladder.
Change of other health-related lifestyles | 6 month and 12 month
  Participants' change of other health-related lifestyles for the drug abuser between baseline, 6-month, 12-month follow-up will use a structured-questionnaire to measure their alcohol consumption, smoking consumption, vegetable and fruit consumption and exercising frequency.
The quality of life | 6 month and 12 month
  Participants' change of quality of life at baseline, 6-month and 12-month follow-up will use EuroQol 5-level scale (EQ-5D-5L) to measure the quality of life. It consists of two part. The first part has 5 questions and each question has choices 1 to 5. Large number means a worse outcome in the first part. The second part has one question which is a scale of 0 to 100. Large number means a better outcome in the second part.
Peer supporters' improvement in professional knowledge towards counselling and treatment | immediately after the training and 6 month
  Peer supporters' improvement in professional knowledge towards counselling and treatment after the training will be measured by a structured questionnaire in pre-training, immediately after the training and 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
The relevant anonymized patient level data, full dataset, technical appendix, and statistical code are available on reasonable request. The approval from the Principal Investigator for the purpose of data use is required.
Time Frame: After the project has been completed and the results of the project has been published
Access Criteria: Request could be sent to Principal Investigator (williamli@cuhk.edu.hk)